CLINICAL TRIAL: NCT03158649
Title: A Novel Web-based Positive Psychology Intervention Addressed to Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Valencia (Other)
Collaborators: University of Twente (Other); Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Rosa María Baños Rivera, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H1429002403332
Record Dates: First submitted 2015-07-02; First posted 2017-05-18 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Pregnancy; Mental Health Wellness 1
Keywords: Pregnancy; Prenatal well-being; Mental maternal prenatal well-being; Positive Psychology; Positive Psychology Intervention; Web-based intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Internet-based Intervention condition (Experimental): Internet-based positive psychology training
  Interventions: Other: "Embarazo y Bienestar"
- Waiting List condition (No Intervention): Waiting List control condition

INTERVENTIONS:
Other: "Embarazo y Bienestar" — The intervention programme is called "Embarazo y Bienestar" ("Pregnancy and Well-being"). Embarazo y Bienestar is a modular, self-placed program mainly designed to foster women's prenatal well-being by practicing some positive psychology-based exercises. The intervention programme consist of four modules of intervention, one welcome module, and a final resume page.
  Arms: Positive Psychology Internet-based Intervention condition

SUMMARY:
The identification and treatment of the disorders connected to the perinatal period has traditionally catalyzed the researchers' attention. Nevertheless, since the World Health Organization has recently coined the concept of positive pregnancy experience, which includes not only treatment of diseases, but also health education, and health promotion, research on antenatal care has expanded to a salutogenic perspective. In the wake of this perspective, a growing number of research have been examining the potential benefits of positive aspects and protective factors on maternal prenatal well-bein. This salutogenic perspective is supported by the emerging field of Positive Psychology. Evidence from Positive Psychology studies has shown that it is possible to build and enhance personal strengths, sense of meaning and positive feelings by practicing some brief positive exercises, called Positive Psychology Interventions (PPIs). Recently, researchers have started to investigate the effects of a PPI on women's prenatal well-being, reporting promising findings in terms of potential direct effects of the positive intervention on women's prenatal stress in comparison to a treatment-as-usual control condition. In the past decade, many web-based delivered interventions have been designed and documented to be effective for the promotion of mental health and for the prevention and treatment of different disorders. Indeed, recent systematic reviews provides preliminary evidence that web-based interventions can be a promising and advisable form of intervention during the perinatal period. PPIs have been translated also in the online format. Preliminary evidence suggests that online positive psychology interventions can effectively enhance well-being and reduce depressive symptoms.

The research team have developed the protocol for a web-based positive psychology programme addressed to promote and enhance women's prenatal well-being. This intervention programme will last five weeks and will be completely self-administered. It is intend to study the effect of the intervention on levels of mental well-being, depression, pregnancy related anxiety and other relevant variables, and the results will be compared to a waiting list control group.

DETAILED DESCRIPTION:
Objective: The aim of this study is to examine the effectiveness of a positive psychology online-based intervention on indices of prenatal wellbeing. Hypotheses: Specifically, the primary hypothesis is that women that would participate to the intervention would report higher levels of mental well-being comparing to the ones reported by women assigned to the control group (i.e., waiting list, WL). Secondly, it is expected that women that would be involve in the positive intervention would report higher levels of positive affect, perceived social support, positive future thinking, and self-acceptance, comparing to the ones reported by the WL group. Moreover it is expected that participants assigned to the intervention condition would report lower levels of negative affect, depression symptoms, pregnancy related anxiety and negative future thinking, comparing to the ones reported by the WL group.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant
* have regular access to Internet
* decided to be the mother of the baby
* Spanish-speaker

Ages: 11 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 164 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Mental well-being | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Warwick-Edinburgh Mental Well-Being Scale (WEMWBS; Tennant et al., 2007)

SECONDARY OUTCOMES:
Changes in Social support | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Multidimensional Scale of Perceived Social Support (MSPSS; Zimet et al., 1988)
Changes in Future directed thinking | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Subjective Probability Task (SPT; MacLeod et al., 1996)
Changes in Affect | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Scale of Positive and Negative Experience (SPANE; Diener et al., 2010)
Changes in Depression | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Patient Health Questionnaire-9 (PHQ-9; Kroenke, & Spitzer, 2002)
Changes in Pregnancy related anxiety | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Pregnancy Related Anxiety Scale (PRAS; Rini et al., 1999)
Changes in Psychological well-being | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Psychological Well-Being Scale (PWBS-29; Ryff, 1989)
Changes in Self-compassion | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Self-Compassion Scale -Short Form (SCS-SF; Raes et al., 2011)
Changes in Satisfaction with life | Baseline, post- training (5-weeks) and at follow-up (5-weeks after post-training)
  Satisfaction With Life Scale (SWLS; Diener, et al., 1985)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Maria Baños, PhD, Study Director — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Background] WHO Recommendations on Antenatal Care for a Positive Pregnancy Experience. Geneva: World Health Organization; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK409108/ PMID 28079998
- [Background] Bos SC, Macedo A, Marques M, Pereira AT, Maia BR, Soares MJ, Valente J, Gomes AA, Azevedo MH. Is positive affect in pregnancy protective of postpartum depression? Braz J Psychiatry. 2013 Mar;35(1):5-12. doi: 10.1016/j.rbp.2011.11.002. PMID 23567594
- [Background] McManus MA, Khalessi AA, Lin J, Ashraf J, Reich SM. Positive feelings during pregnancy, early feeding practices, and infant health. Pediatr Int. 2017 May;59(5):593-599. doi: 10.1111/ped.13209. Epub 2017 Feb 14. PMID 27914182
- [Background] Voellmin A, Entringer S, Moog N, Wadhwa PD, Buss C. Maternal positive affect over the course of pregnancy is associated with the length of gestation and reduced risk of preterm delivery. J Psychosom Res. 2013 Oct;75(4):336-40. doi: 10.1016/j.jpsychores.2013.06.031. Epub 2013 Jul 9. PMID 24119939
- [Background] Seligman ME, Steen TA, Park N, Peterson C. Positive psychology progress: empirical validation of interventions. Am Psychol. 2005 Jul-Aug;60(5):410-21. doi: 10.1037/0003-066X.60.5.410. PMID 16045394
- [Background] Matvienko-Sikar K, Dockray S. Effects of a novel positive psychological intervention on prenatal stress and well-being: A pilot randomised controlled trial. Women Birth. 2017 Apr;30(2):e111-e118. doi: 10.1016/j.wombi.2016.10.003. Epub 2016 Oct 31. PMID 27810284
- [Background] Ashford MT, Olander EK, Ayers S. Computer- or web-based interventions for perinatal mental health: A systematic review. J Affect Disord. 2016 Jun;197:134-46. doi: 10.1016/j.jad.2016.02.057. Epub 2016 Mar 9. PMID 26991368
- [Background] Lee EW, Denison FC, Hor K, Reynolds RM. Web-based interventions for prevention and treatment of perinatal mood disorders: a systematic review. BMC Pregnancy Childbirth. 2016 Feb 29;16:38. doi: 10.1186/s12884-016-0831-1. PMID 26928898
- [Background] Bolier L, Abello KM. Online positive psychological interventions: State of the art and future directions. In Parks AC, Schueller SM editors. The Wiley Blackwell handbook of positive psychological interventions. Chichester, UK: John Wiley & Sons, Ltd; 2014. p. 286-309.